CLINICAL TRIAL: NCT06874036
Title: Safety, Efficacy and Tolerability of Bowel Preparation and Colonoscopy in Patient With Chronic Heart Disease, Chronic Kidney Disease and Chronic Liver Disease
Brief Title: Safety, Efficacy and Tolerability of Bowel Preparation and Colonoscopy in Patient With CHD, CKD and CLD
Status: Recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Director, Asian Institute of Gastroenterology, India
Other Study IDs: Bowel01
Record Dates: First submitted 2025-02-22; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Colon Disease
MeSH Terms: conditions — Colonic Diseases | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Colonoscopy — Colonoscopy is a procedure to see the ascending, transverse, decending, sigmoid, rectum of colon parts

SUMMARY:
Consecutive eligible patients will be enrolled and written informed consent will be obtained from all participants. Routine blood investigations will be sent. Patients with chronic heart failure will be classified based on ejection fraction into 2 groups (EF </> 40%), patients with chronic kidney disease will be classified based on KDIGO classification system into grade I-V. Patients with chronic liver disease will be classified according to the child pugh scoring system into three groups (Child A, B and C). All patients will be undergo bowel preparation under supervision. The patients will be given 10 mg of bisacodyl, the night before colonoscopy. A PEG sachet (137.15 g) containing polyethylene glycol (118 g), sodium chloride (2.93 g), potassium chloride (1.484 g), sodium bicarbonate (3.370 g), and anhydrous sodium sulfate (11.36 g) will be constituted into 2 L solution and used for bowel preparation.

Patients will receive 1 L of PEG solution between 10 PM and 11 PM the day before and 1 L of PEG solution between 6 AM and 7 AM on the day of colonoscopy. Clear liquids will be allowed after the completion of the last bowel preparation until the start of the procedure. Liquid diet includes soups, fruit juices, rice kanji, or porridge in liquid consistency, and clear liquids such as coconut water and lemon juice.

After the adequacy of bowel preparation is deemed fit, the patients will be taken for colonoscopic examination. A single blinded outcome assessment will be done by the colonoscopist/endoscopist performing the procedure (adequacy of bowel preparation) and the endoscopy nurse (tolerability and compliance).

Colonoscopy will be performed using standard video colonoscopes (Olympus, Tokyo, Japan) between 11:00 AM and 1:00 PM without sedation. The colonoscopist / endoscopist will assess the adequacy of bowel preparation using the Boston Bowel Preparation Scale (BBPS). Excellent, good and poor bowel preparations will be defined by BBPS score of 9, 6 - 9 and < 6, respectively. (12-14) Blood sampling will be done before bowel preparation and after colonoscopy in all patients for measurement of baseline parameters, renal function status (Serum creatinine, serum urea), serum electrolytess (serum sodium, serum potassium, serum phosphate and serum calcium) and haematocrit.

Assessment of safety and tolerability will be performed using clinical examination and symptom questionnaire. Cardiovascular and gastrointestinal (GI) symptoms will be recorded. Cardiovascular symptoms such as dyspnea, palpitations, chest pain, will be recorded and scored using the NYHA classification system for symptom severity. Clinical examination will be carried out post-bowel preparation and post-procedure to assess for signs of fluid overload, i.e. auscultation for crepitations and measurement of JVP. GI symptoms such as nausea, abdominal pain, vomiting, dizziness, bloating, and headache will be recorded and scored on a 4-point scale: 1 = none, 2 = mild, 3 = moderate, and 4 = severe. The compliance of bowel preparation will be defined as "poor" for patients who consume less than 75% of the PEG preparation.

DETAILED DESCRIPTION:
Primary objective

• Safety of split dose 2 litre PEG bowel preparation in patients with underlying chronic conditions

Secondary objective

* Adequacy of bowel preparation using Boston bowel preparation scale
* Compliance of bowel preparation
* Change from baseline to post-procedural JVP
* Percentage of patients requiring hospitalization post-procedure

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years
* Diagnosed cases of chronic heart disease, chronic kidney disease or chronic liver failure planned for elective colonoscopy

Exclusion Criteria:

* Age < 18 years
* Current or past history of bowel obstruction or resection
* Known allergies to PEG
* Emergency colonoscopies.
* Pregnant or lactating women
* Paralytic ileus / Bowel perforation
* Inability to protect airway

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 74 subjects
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
To check the large intestine | 60 minutes
  to clear the contents in intestine like faces in gm/dl

CONTACTS AND LOCATIONS:
Overall Officials: Manohar Dr Reddy, MBBS MD, Principal Investigator — AIG Hospitals
Locations (1):
- Asian Institute of Gastroenterology/AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No